CLINICAL TRIAL: NCT00372892
Title: A Randomized, Double Blind, Placebo Controlled Pilot Trial of Rituximab for Non-splenectomized Adults With Acute Immune Thrombocytopenic Purpura Receiving Standard Treatment (R-ITP)
Brief Title: Pilot Study of Rituximab for the Treatment of Acute Immune Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Donald Arnold, MD, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-105; HC-104634
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: Idiopathic Thrombocytopenic Purpura; Rituximab; Feasibility study
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Rituximab
  Interventions: Drug: Rituximab
- B (Placebo Comparator): Saline placebo iv infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — 375mg/m2 per week for 4 consecutive weeks
  Other Names: Rituxan, Mabthera
  Arms: A
Drug: Placebo — Saline IV placebo once per week for 4 consecutive weeks
  Arms: B

SUMMARY:
The purpose of this study is to assess the feasibility of a randomized, double blind, placebo controlled trial of add-on rituximab for non-splenectomized adults with acute immune thrombocytopenic purpura (ITP).

DETAILED DESCRIPTION:
Immune thrombocytopenic purpura (ITP) is an autoimmune disease characterized by severe thrombocytopenia and bleeding. With current standard therapies, adult-onset ITP tends to recur thus exposing patients to prolonged risks of hemorrhage and toxicities of standard treatments. Rituximab, a chimeric anti-CD20 monoclonal antibody, has been shown to be effectively raise the platelet count in some patients with ITP and there is clinical and biological evidence to suggest that, if given early, rituximab may prevent ITP relapses.

We have designed a randomized, double blind, placebo controlled pilot trial of rituximab for the treatment of non-splenectomized adults with acute ITP who are receiving standard treatments. The primary objectives of this trial are to determine the feasibility of recruitment, randomization and blinding; the safety of rituximab in ITP; and the event rate in the control group which will be used to calculate the sample size for a larger trial. Secondary objectives are to determine rates of 6-month event free survival where an event is defined as any of: a platelet count <50; the need for rescue treatment; or significant bleeding. Data from this pilot trial will inform the design of a larger phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Non-splenectomized patients with acute ITP, where "acute ITP" is defined as a platelet count below 30 at the time that standard treatment was recommended by a physician and for which no treatment had been received for the preceding 30 days.
* Must be receiving standard ITP treatment.

Exclusion Criteria:

* Cardiac arrhythmia.
* Uncontrolled hypertension or inability to hold antihypertensive medications for 12 hours prior to and throughout study drug infusions.
* Known coronary artery disease, angina pectoris or myocardial infarction within the last year.
* Significant pulmonary disease within the last year.
* Stroke, transient ischemic attack or venous thrombosis within the last year.
* Secondary causes of thrombocytopenia (splenomegaly [palpable spleen or radiologically confirmed >14 cm], drug-induced thrombocytopenia, hereditary thrombocytopenia, microangiopathic hemolytic anemia, myelodysplastic syndrome).
* Chronic lymphocytic leukemia or lymphoma.
* Active or metastatic cancer.
* History of hepatitis B or C or HIV.
* Active infection in the 4 weeks before randomization.
* Inherited coagulation factor deficiency.
* Aspirin, aspirin-containing compounds, salicylates, non-steroidal anti-inflammatory medications (NSAIDS) medications, clopidogrel or ticlopidine in the 7 days preceding study drug infusions; vitamin K antagonists (warfarin) in the 3 days preceding study drug infusions; unfractionated heparin or low molecular weight heparin in the 24 hours preceding study drug infusions.
* Elevated INR or prolonged PTT; LDH, serum creatinine, liver function tests (AST/SGOT, ALT/SGPT, alkaline phosphatase, total bilirubin) increased more than 1.5 times upper limit of normal.
* Prior rituximab treatment.
* Unable to schedule 4 weekly study infusions.
* Pregnancy or breastfeeding.
* Known sensitivity to murine proteins, Chinese Hamster Ovary (CHO) cell proteins or to any component of rituximab.
* Participation in another clinical trial.
* Geographic inaccessibility.
* Failure to provide written informed consent.
* Any additional laboratory test result, health related illness or other diagnosis which, in the opinion of the treating physician, may put the subject's health or safety at risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | 3 years
Degree of adherence to the study protocol | 3 years
Event free survival in controls | 6 months
Bleeding | 6 months
rescue therapy | 6 months

SECONDARY OUTCOMES:
Platelet count response | 6 months
Quality of life | 6 months
Circulating CD-20 positive lymphocytes | 6 months
Platelet associated IgG | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Arnold, MD, Principal Investigator — McMaster University
Locations (7):
- Canada (7):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster Univerisity, Hamilton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Arnold DM, Heddle NM, Carruthers J, Cook DJ, Crowther MA, Meyer RM, Liu Y, Cook RJ, McLeod A, MacEachern JA, Mangel J, Anderson D, Vickars L, Tinmouth A, Schuh AC, Kelton JG. A pilot randomized trial of adjuvant rituximab or placebo for nonsplenectomized patients with immune thrombocytopenia. Blood. 2012 Feb 9;119(6):1356-62. doi: 10.1182/blood-2011-08-374777. Epub 2012 Jan 5. PMID 22223819
- [Derived] Arnold DM, Crowther MA, Meyer RM, Carruthers J, Ditomasso J, Heddle NM, McLeod A, Kelton JG. Misleading hepatitis B test results due to intravenous immunoglobulin administration: implications for a clinical trial of rituximab in immune thrombocytopenia. Transfusion. 2010 Dec;50(12):2577-81. doi: 10.1111/j.1537-2995.2010.02766.x. PMID 20576011